CLINICAL TRIAL: NCT03322332
Title: The Role of Adipokines Secreted by Epicardial Adipose Tissue in the Atherosclerosis of Coronary Arteries
Brief Title: Adipokines of Epicardial Adipose Tissue and Atherosclerosis of Coronary Arteries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Georgios A. Christou, Cardiologist, Postdoctoral researcher, University Hospital, Ioannina
Other Study IDs: 741
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Coronary Atherosclerosis; Adipokines
Keywords: adiponectin; omentin-1; resistin; RBP4; epicardial fat; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- NonDM-0: Nondiabetics without significant stenoses (> 50%) in the coronary arteries
- NonDM-L: Nondiabetics with significant stenosis in the left anterior descending (LAD) coronary artery or in the Left main (LM) coronary artery, but without significant stenosis in the right coronary artery (RCA)
- NonDM-R: Nondiabetics without significant stenosis in the LAD and in the LM, but with significant stenosis in the RCA
- NonDM-LR: Nondiabetics with significant stenosis in the LAD or in the LM and with significant stenosis in the RCA
- DM-0: Patients with type 2 diabetes mellitus (T2DM) without significant stenoses in the coronary arteries
- DM-L: T2DM patients with significant stenosis in the LAD or in the LM, but without significant stenosis in RCA
- DM-R: T2DM patients without significant stenosis in the LAD and in the LM, but with significant stenosis in the RCA
- DM-LR: T2DM patients with significant stenosis in the LAD or in the LM and with significant stenosis in the RCA

SUMMARY:
The aim of the study is to investigate whether the expression and production of adipokines secreted by the epicardial adipose tissue correlate with the degree of coronary atherosclerosis.

DETAILED DESCRIPTION:
The aim of the study is to investigate whether the expression and production of four adipokines [adiponectin, omenin-1, resistin and retinol binding protein-4 (RBP4)] secreted by the epicardial adipose tissue correlate with the degree of coronary atherosclerosis. Specifically, this study aims to investigate whether the expression and production of these adipokines is different between two sites of the heart, that are perfused by coronary arteries with different degrees of stenosis.

ELIGIBILITY:
Inclusion Criteria:

1) Individuals undergoing cardiac surgery

Exclusion Criteria:

* Age < 18 years
* HbA1c > 7.0%
* Any change of antidiabetic medication the previous 3 months before the surgery
* GFR < 60 mL/min/1.73 m2
* Liver disease
* Cancer
* Non-treated hyperthyroidism or hypothyroidism
* Autoimmune disease
* Infection
* Any change in body weight at least 5% the previous 3 months before surgery
* Significant dehydration.
* Taking any of the following drugs the previous 3 months before surgery: hormones, antiobesity drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals undergoing cardiac surgery will be recruited in this study.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-01-15 (Estimated); Study Completion 2018-01-22 (Estimated)

PRIMARY OUTCOMES:
Association between coronary artery disease and epicardial adipokines | Baseline measurement
  Comparison of the mRNA and protein production of four adipokines [adiponectin, omentin-1, resistin, retinol binding protein-4(RBP4)] from the epicardial adipose tissue between the territories that are supplied by LAD and RCA. This comparison will be performed in the following clusters of groups:
  1. Cluster 1: NonDM-0 and DM-0 (comparison between territories that are supplied by non-stenosed coronary arteries)
  2. Cluster 2: NonDM-LR and DM-LR (comparison between territories that are supplied by stenosed coronary arteries)
  3. Cluster 3: NonDM-L, NonDM-R, DM-L and DM-R (comparison between a territory that is supplied by stenosed coronary artery and another territory that is supplied by non-stenosed coronary artery)

SECONDARY OUTCOMES:
Impact of diabetes on epicardial adipokines | Baseline measurement
  Comparison of the mRNA and protein production of four adipokines (adiponectin, omentin-1, resistin, RBP4) from the epicardial adipose tissue of the territory that is supplied by LAD or RCA between the following groups:
  1. NonDM-0 vs DM-0
  2. NonDM-L vs DM-L
  3. NonDM-R vs DM-R
  4. NonDM-LR vs DM-LR

CONTACTS AND LOCATIONS:
Overall Officials: Eustratios Apostolakis, Professor, Study Director — University Hospital, Ioannina
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece